CLINICAL TRIAL: NCT03559686
Title: Named Patient Program With Certolizumab Pegol in Adults Suffering From Rheumatoid Arthritis (RA) Who Participated in Open Label Studies C87015, C87028 and C87051
Brief Title: Named Patient Program With Certolizumab Pegol in Adults Suffering From Rheumatoid Aarthritis (RA)
Status: Available | Type: Expanded Access
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: RA0039
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Certolizumab Pegol — The recommended maintenance dose of Cimzia® (Certolizumab Pegol) for adult patients with Rheumatoid Arthritis (RA) is 200 mg every 2 weeks (single 1 mL injection of 200 mg) .
  Other Names: Cimzia

SUMMARY:
The objective of this Named Patient Program (NPP) is to provide continued availability of Certolizumab Pegol (CZP) to adult Rheumatoid Arthritis (RA) patients who participated in the open label studies C87015 (CDP870 015), C87028 (CDP870-028) and C87051 (CDP870-051). Physicians may use the option to continue offering patients CZP treatment or to transition patients off CZP to a standard care regimen.

ELIGIBILITY:
Inclusion Criteria:

* Has/will complete(d) one of the Certolizumab Pegol (CZP) open-label studies (C87015, C87028, C87051)
* Is currently taking CZP (last dose within the last 6 weeks for subjects from C87015, and within the last 4 weeks for subjects from C87028 or C87051)
* Is informed of the details of this Named Patient Program (NPP), is given ample time and opportunity to ask questions in order to consider his/her participation in this NPP and has provided verbal consent to participate, and, if applicable according to local regulations, has given his/her written informed consent for participation

Exclusion Criteria:

* Has been treated with any experimental biological or nonbiological therapy other than CZP within 5 plasma half-lives
* Current safety concerns for continuing an CZP therapy related to prior biologic therapy (eg, insufficient wash out period, unresolved adverse events, unresolved recovery of peripheral B-cell/lymphocyte levels following therapy with B-cell depleters)
* Has received live vaccinations including, but not limited to, oral polio, herpes zoster, measles-mumps-rubella (MMR) or nasal influenza within the last 8 weeks or has planned live immunizations during the planned period of administration of CZP
* Serious or life-threatening infection within the last 6 months, including any herpes zoster infection, and/or any signs of current or recent infection
* Active or latent tuberculosis (TB): if one or more of the 3 criteria is positive for evidence of TB infection:

  1. A medical history of or current active tuberculosis (TB)
  2. A recent (<6 months) chest X-ray with signs consistent with TB infection
  3. A recent (<6 months) positive purified protein derivative (PPD) skin test (defined as induration or 5 mm or more) and/or an indeterminate or positive QuantiFERON-TB Gold or Elispot test.

Patients must be monitored at least annually for active and latent TB by both 1) a chest X-ray read by a pulmonologist or radiologist and 2) a PPD skin test and/or Elispot/ QuantiFERON TB Gold test.

* Concurrent known acute or chronic viral hepatitis B or C infection
* Concurrent known human immunodeficiency virus (HIV) infection
* Concurrent malignancy or a history of malignant disease
* History of a lymphoproliferative disorder or any signs or symptoms suggestive of this disease
* History of, or suspected or confirmed active demyelinating disease of the central nervous system
* History of or concurrent New York Heart Association (NYHA) Class III/IV heart failure
* Current or recent history of severe, progressive, uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)